CLINICAL TRIAL: NCT05073523
Title: Dietary Biomarkers 2.0: From Potential Towards Implementation. A Randomized Controlled Trial to Assess Dose-response Relationships for Dietary Biomarkers of Selected Foods
Brief Title: Dietary Biomarkers 2.0: From Potential Towards Implementation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Responsible Party: Principal Investigator, Rikard Landberg, Professor, Chalmers University of Technology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: ChalmersUT
Record Dates: First submitted 2021-09-06; First posted 2021-10-11 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Healthy
MeSH Terms: interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meal A (Other): Diet: meal proportion 1
  Interventions: Other: Diet
- Meal B (Other): Diet: meal proportion 2
  Interventions: Other: Diet
- Meal C (Other): Diet: meal proportion 3
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — All intervention meals consist of five different food groups including fruits, vegetables, legumes, dairy products, and whole grains. Differences in the proportion of these foods in Meal A-C is tested.

SUMMARY:
The aim of this project is to fill a gap in the translation of dietary biomarkers as unbiased measures of food intake from high-end academic research into a methodology that ca be easily applied across academic, public and private health sector to objectively assess specific dietary intakes at group and individuals' level to a) improve understanding of diet and health relationships b) address compliance in dietary intervention studies and c) assess individuals' dietary intakes to guide their eating towards improved health. The study will be carried out as a three-way cross-over design with three different meal compositions (A, B, C) where each meal is provided 3 times per day during four days per meal. A wash-out period of 7 days where participants consume their habitual diet is implemented and a 3-day run-in before the study meal intervention. The first day of study meal intervention includes postprandial measurements during 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 18-80 years
* Body mass index (BMI) 18.5-30 kg/m2
* Fasting glucose ≤ 6.1 mmol/l
* Low density lipoprotein (LDL), Cholesterol ≤ 5.30 mmol/L
* Triglycerides ≤ 2.60 mmol/L
* Signed informed consent

Exclusion Criteria:

* Food allergies or intolerances preventing consumption of any products included in the study.
* Strict vegetarian or vegan, participants must be able to eat dairy products as it is included in the study diet.
* Unable to sufficiently understand written and spoken Swedish to provide written consent and understand information and instructions from the study personal.
* Unable to satisfactorily complete the 3-day weighted food records.
* Continuous/daily use of medication.
* Pregnant, lactating or planning a pregnancy during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of dietary candidate biomarkers (daidzein, genistein, hesperetin, naringenin, phloretin, kaempferol, 2-thiothiazolidine-4-carboxylic acid, sulforaphane) | 24 hours
  Difference in the plasma concentrations of diet specific biomarkers comparing before (baseline) and after intervention meal (average plasma concentration over the 24h period).
Plasma concentrations of dietary biomarker candidates (proline betaine, 4-hydroxyphenylacetic acid, 4-hydroxyphenylpyruvate, indole-3-lactic acid, pipecolic acid, s-methylcysteine, avenacoside-A and avenacoside-B) | 24 hours
  Difference in the plasma concentrations of diet specific biomarkers comparing before (baseline) and after intervention meal (average plasma concentration over the 24 h period).
Plasma concentration-time profile over 24h (AUCs) of dietary biomarker candidates ( daidzein, genistein, hesperetin, naringenin, phloretin, kaempferol, 2-thiothiazolidine-4-carboxylic acid, sulforaphane) | 24 hours
  Differences in plasma AUCs between the three intake levels for each biomarker candidate
Plasma concentration-time profile over 24h (AUCs) of dietary biomarker candidates proline betaine, 4-hydroxyphenylacetic acid, 4-hydroxyphenylpyruvate, indole-3-lactic acid, pipecolic acid, s-methylcysteine, avenacoside-A and avenacoside-B | 24 hours
  Differences in plasma AUCs between the three intake levels.

SECONDARY OUTCOMES:
Gut microbiome | 4 days
  Fecal samples will analyzed for composition of the gut microbiome, baseline compared with after 4 days of intervention meals.
Plasma metabolites | 4 days
  Untargeted metabolomics will be performed using established methods for plasma. Analyzed exploratorily using untargeted metabolomics to find potential biomarker panels that reflect the specific foods included in study meals. Baseline compared with after intervention meals.
Urine metabolites | 24 hours
  Analyzed exploratorily using untargeted metabolomics to find potential biomarker panels that reflect the specific foods included in study meals.
Fecal concentrations of diet specific biomarkers daidzein, genistein, hesperetin, naringenin, phloretin, kaempferol, 2-thiothiazolidine-4-carboxylic acid, sulforaphane | 4 days
  Evaluate new simple sampling techniques using faecal swabs.
Fecal concentrations of diet specific biomarkers proline betaine, 4-hydroxyphenylacetic acid, 4-hydroxyphenylpyruvate, indole-3-lactic acid, pipecolic acid, s-methylcysteine, avenacoside-A and avenacoside-B) | 4 days
  Evaluate new simple sampling techniques using fecal swabs.
Blood concentrations of diet specific biomarkers daidzein, genistein, hesperetin, naringenin, phloretin, kaempferol, 2-thiothiazolidine-4-carboxylic acid, sulforaphane | 4 days
  Evaluate new simple sampling techniques using dried blood spots.
Blood concentrations of diet specific biomarkers proline betaine, 4-hydroxyphenylacetic acid, 4-hydroxyphenylpyruvate, indole-3-lactic acid, pipecolic acid, s-methylcysteine, avenacoside-A and avenacoside-B) | 4 days
  Evaluate new simple sampling techniques using dried blood spots.
Urine concentrations of diet specific biomarkers daidzein, genistein, hesperetin, naringenin, phloretin, kaempferol, 2-thiothiazolidine-4-carboxylic acid, sulforaphane | 4 days
  Evaluate new simple sampling techniques using dried urine spots.
Blood concentrations of diet specific biomarkers proline betaine, 4-hydroxyphenylacetic acid, 4-hydroxyphenylpyruvate, indole-3-lactic acid, pipecolic acid, s-methylcysteine, avenacoside-A and avenacoside-B | 4 days
  Evaluate new simple sampling techniques using dried urine spots.

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Landberg, Dr, Principal Investigator — Chalmers University of Technology
Locations (1):
- University of Gothenburg, Department of Food and Nutrition and Sport Science, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No